CLINICAL TRIAL: NCT05732844
Title: Efficacy of the Use of Vaginal Balls for the Improvement of Urinary Incontinence and Sexual Function in Women. Randomized Control Trial.
Brief Title: Efficacy of the Use of Vaginal Balls for the Improvement of Urinary Incontinence and Sexual Function in Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAPbarcelona (Other)
Responsible Party: Principal Investigator, Inés Ramírez-García, Director, RAPbarcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAIA_bolas
Record Dates: First submitted 2023-01-29; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Urinary Incontinence; Stress Urinary Incontinence; Sexual Dysfunction
Keywords: vaginal spheres; physiotherapy; pelvic floor muscle trainning
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress; Sexual Dysfunction, Physiological | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group with Enna pelvic ball (Experimental): This group will receive instructions on how to carry out PFMT daily at home, and indications for the placement of Enna pelvic ball vaginal spheres daily.
  Interventions: Device: Intervention group with Enna pelvic ball
- Control group (Active Comparator): This group will receive instructions on how to carry out PFMT daily at home.
  Interventions: Other: Control group

INTERVENTIONS:
Device: Intervention group with Enna pelvic ball — The home guideline for placement of the vaginal spheres will be as described in next:
  st-2nd week 15 minutes, 1 time a day nd-4th week 30 minutes, 1 time a day 4th-8th week 1 hour, 1 time a day 8th-12th week 2 hours, 1 time a day 12th-16th week 3 hours, 1 time a day
  Arms: Intervention group with Enna pelvic ball
Other: Control group — According to the PERFECT score, a daily home guideline for the performance of PFMT will be requested three times a day, two types of exercises (endurance and strength), and eight repetitions of each.
  Arms: Control group

SUMMARY:
Asess if adding vaginal spheres treatment to the conventional Pelvic Floor Muscle Trainning (PFMT) produces a greater decrease in the severity of the stress urinary incontinence or a greater perceived quality of life related to incontinence.

DETAILED DESCRIPTION:
The intervention group will perform the pelvic floor muscle trainning (PFMT) plus the use of vaginal spheres, while the control group will perform the PFMT treatment only, daily at home. The study will be conducted on women with stress urinary incontinence. The intervention will last four months and will consist of a monthly session with the physiotherapist, doing a total of 4 sessions and the final assessment.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 or over
* Suffer from stress urinary incontinence or mixed urinary incontinence.
* Understand Spanish to be able to self-complete the questionnaires (validated in Spanish).

Exclusion Criteria:

* Not giving informed consent.
* Women with faecal incontinence.
* Women with grade III-IV prolapse.
* Women with pathology that can affect the neuro-muscular response.
* Women with incontinence that is not of functional origin.
* Women who have perineal pain that makes it impossible to apply the spheres.
* Women with an open vagina of more than 2.5 cm opening
* Being pregnant.
* Not being committed to complying with a minimum of 80% of the treatment.
* Having previously started other pelvic physiotherapy treatments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Severity of urinary incontinence using the ICIQ-SF questionnaire (International Consultation on Incontinence Questionnaire Short form) at Week 16. | Time Frame: Baseline and Week 16
  The ICIQ-SF is a validated self-reported instrument assessing the urinary incontinence severity and It's quality of life. Possible scores range from 0 (no incontinence) to 21 (severe incontinence). Change=(Week 16 score - baseline score).

CONTACTS AND LOCATIONS:
Locations (1):
- RAPbarcelona SL, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Oblasser C, Christie J, McCourt C. Vaginal cones or balls to improve pelvic floor muscle performance and urinary continence in women post partum: A quantitative systematic review. Midwifery. 2015 Nov;31(11):1017-25. doi: 10.1016/j.midw.2015.08.011. Epub 2015 Sep 9. PMID 26428191